CLINICAL TRIAL: NCT05677893
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Inhaled MBS-COV (SNS812) in Healthy Participants
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Inhaled MBS-COV (SNS812) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SNS812CLCT01
Record Dates: First submitted 2022-11-04; First posted 2023-01-10 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Disease Caused by Severe Acute Respiratory Syndrome Coronavirus 2 (Disorder)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational drug (Experimental): Eligible participants will be assigned to receive 0.3-1.2 mg/kg single or multiple doses of the investigational drug.
  Interventions: Drug: MBS-COV
- Placebo (Placebo Comparator): Eligible participants will be assigned to single or multiple doses of the placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MBS-COV — MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
  Arms: Investigational drug
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Inhaled MBS-COV in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive).
* No serious or chronic underlying disease which would adversely affect the study conduct and data interpretation per the investigator.
* Female participants should have negative results in serum pregnancy test at screening and negative urine pregnancy test at admission
* Participants with normal spirometry (FEV1: 90% or greater) results at screening or day -1.
* Both male and female participants and their partners of childbearing potential must agree to use two medically accepted methods of contraception.
* Participants should have normal (or abnormal but not clinically significant) laboratory results per the PI's judgement including the hematology, biochemistry, coagulation indices, and urinalysis.
* Participants should have a normal (or abnormal but not clinically significant) 12-lead ECG at screening and day -1 and chest X-ray at screening
* Participants should be willing to cooperate and able to participate in this study, comply with all protocol requirements, and sign an informed consent.
* Current non-smokers and those who have not smoked within the last 3 months. This includes the use of cigarettes, e-cigarettes, and nicotine replacement products.
* Nasopharyngeal or nasal swab sample of Participants collected for COVID-19 antigen rapid test at screening and qRT-PCR test on Day -1 should be negative.

Exclusion Criteria:

* The participant has a known history of, or a positive test result for, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at screening.
* As reported by the participant has severe cardiovascular disease, neurological disease, hematological disease, infectious disease, mental disorder, liver disease, gastrointestinal disease, lung disease, endocrine disease, immune disease or kidney disease, or has a history of the above diseases, or other symptoms known to interfere with the absorption, distribution, metabolism, or excretion of the medicine, or other conditions that the investigator believes will increase the risk of the participant and might interfere with the study conduct and results interpretation.
* The participant has history or presence of active lung disease (i.e., asthma, chronic obstructive pulmonary disease [COPD], pulmonary fibrosis, hemoptysis, bronchiectasis) or prior intubation.
* The participant has upper respiratory infection within the 3 months prior to the first dose of study drug.
* Consumed more than 14 units of alcohol per week in the 6 months before screening (1 unit of alcohol = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) or have taken alcohol products in the 48 hours prior to administration, or those who have a positive alcohol breath test result at screening and day -1.
* Unwillingness to abstain from the consumption of any caffeine or alcohol-containing food or drinks that may influence the drug metabolism from 48 hours before administration.
* History of drug abuse or a positive drug abuse (barbiturates, methamphetamine, benzodiazepines, morphine/opiates, phencyclidine (PCP), amphetamines, tetrahydrocannabinol (THC), methylenedioxymethamphetamine (MDMA), cocaine, methadone, and cotinine) test result at screening and day -1.
* Female participants who are lactating.
* Use of prescription or non-prescription drugs, including vaccine within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
* The subject has received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month prior to the first dose of study drug and will receive another experimental agent during the duration of this study.
* The participant has a history of frequent nose bleeding.
* Participants with known allergic reactions to the study drug or its excipients.
* The participant has an acute sinusitis or history of chronic sinusitis, a history of active allergic rhinitis (AR), history of perennial allergic rhinitis (PAR), or current seasonal allergic rhinitis (SAR), or recent viral rhinitis within 2 weeks prior to administration.
* The participant has Any nasopharyngeal abnormality that may have interfered with nasal absorption, distribution, or study-related evaluations of signs or symptoms (e.g., polyps, septal deviation).
* Blood donation of more than 400 mL within 3 months before screening or more than 200 mL within 4 weeks before screening or plan to donate blood during study period.
* Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Unit, Los Angeles, California, United States

REFERENCES:
- [Derived] Chang YC, Chen YF, Yang CF, Ho HJ, Yang JF, Chou YL, Lin CW, Yang PC. Pharmacokinetics and Safety Profile of SNS812, a First in Human Fully Modified siRNA Targeting Wide-Spectrum SARS-CoV-2, in Healthy Subjects. Clin Transl Sci. 2025 Mar;18(3):e70202. doi: 10.1111/cts.70202. PMID 40116355

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Drug, 0.3 mg/kg, Part A (SAD): Eligible participants will be assigned to receive a 0.3 mg/kg single dose of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Investigational Drug, 0.6 mg/kg, Part A (SAD): Eligible participants will be assigned to receive a 0.6 mg/kg single dose of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Investigational Drug, 1.2 mg/kg, Part A (SAD): Eligible participants will be assigned to receive a 1.2 mg/kg single dose of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Placebo, Part A (SAD): Eligible participants will be assigned to single doses of the placebo. Placebo: Normal saline
- Investigational Drug, 0.6 mg/kg, Part B (MAD): Eligible participants will be assigned to receive 0.6 mg/kg multiple doses of the investigational drug, once daily for 7 consecutive days.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Investigational Drug, 1.2 mg/kg, Part B (MAD): Eligible participants will be assigned to receive 1.2 mg/kg multiple doses of the investigational drug, once daily for 7 consecutive days.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Placebo, Part B (MAD): Eligible participants will be assigned to multiple doses of the placebo, once daily for 7 consecutive days.
  Placebo: Normal saline
Period: Overall Study
Arm/Group | Investigational Drug, 0.3 mg/kg, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part A (SAD) | Investigational Drug, 1.2 mg/kg, Part A (SAD) | Placebo, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part B (MAD) | Investigational Drug, 1.2 mg/kg, Part B (MAD) | Placebo, Part B (MAD)
Started | 6 | 6 | 6 | 6 | 8 | 8 | 4
Completed | 5 | 6 | 6 | 6 | 7 | 7 | 4
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Others | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Investigational Drug, 0.3 mg/kg, Part A (SAD): Eligible participants will be assigned to receive 0.3 mg/kg single doses of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Investigational Drug, 0.6 mg/kg, Part A (SAD): Eligible participants will be assigned to receive 0.6 mg/kg single doses of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Investigational Drug, 1.2 mg/kg, Part A (SAD): Eligible participants will be assigned to receive 1.2 mg/kg single doses of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Investigational Drug, 0.6 mg/kg, Part B (MAD); Investigational Drug, 1.2 mg/kg, Part B (MAD): Eligible participants will be assigned to receive 0.6 mg/kg mutiple doses of the investigational drug.
  MBS-COV: MBS-COV is a potent siRNA treatment for mild to moderate COVID-19.
- Placebo, Part B (MAD): Eligible participants will be assigned to multiple doses of the placebo.
  Placebo: Normal saline
- Total: Total of all reporting groups
Arm/Group | Investigational Drug, 0.3 mg/kg, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part A (SAD) | Investigational Drug, 1.2 mg/kg, Part A (SAD) | Placebo, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part B (MAD) | Investigational Drug, 1.2 mg/kg, Part B (MAD) | Placebo, Part B (MAD) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 4 | 44
Age, Customized [Mean (Standard Deviation); unit: years] | 37.67 (9.09) | 38.83 (7.47) | 30.83 (6.8) | 31.83 (10.5) | 35.13 (5.38) | 36.38 (9.61) | 37.5 (8.89) | 36.1 (7.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 0 | 2 | 4 | 0 | 12
  Male | 5 | 5 | 2 | 6 | 6 | 4 | 4 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 1 | 1 | 2 | 1 | 12
  Not Hispanic or Latino | 5 | 3 | 3 | 5 | 7 | 6 | 3 | 32
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 8 | 8 | 4 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by Protocol Definition of AE
Description: Safety will be reported based on Protocol defined AEs.
  For the purpose of this protocol, an AE will be defined as any untoward medical occurrence in a subject during the study.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- Investigational Drug, 0.3 mg/kg, Part A (SAD): Eligible participants will be assigned to receive 0.3 mg/kg single doses of the investigational drug.
- Investigational Drug, 0.6 mg/kg, Part A (SAD): Eligible participants will be assigned to receive 0.6 mg/kg single doses of the investigational drug.
- Investigational Drug, 1.2 mg/kg, Part A (SAD): Eligible participants will be assigned to receive 1.2 mg/kg single doses of the investigational drug.
- Placebo, Part A (SAD): Eligible participants will be assigned to single doses of the placebo.
- Investigational Drug, 0.6 mg/kg, Part B (MAD); Investigational Drug, 1.2 mg/kg, Part B (MAD): Eligible participants will be assigned to receive 0.6 mg/kg mutiple doses of the investigational drug.
Arm/Group | Investigational Drug, 0.3 mg/kg, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part A (SAD) | Investigational Drug, 1.2 mg/kg, Part A (SAD) | Placebo, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part B (MAD) | Investigational Drug, 1.2 mg/kg, Part B (MAD) | Placebo, Part B (MAD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 4
Participants | 3 | 0 | 0 | 1 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: From start of treament on Day 1 to Day 28
Groups:
- Placebo, Part B (MAD): Eligible participants will be assigned to multiple doses of the placebo.
Arm/Group | Investigational Drug, 0.3 mg/kg, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part A (SAD) | Investigational Drug, 1.2 mg/kg, Part A (SAD) | Placebo, Part A (SAD) | Investigational Drug, 0.6 mg/kg, Part B (MAD) | Investigational Drug, 1.2 mg/kg, Part B (MAD) | Placebo, Part B (MAD)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6 | 0/6 | 1/6 | 0/8 | 2/8 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Drug, 0.3 mg/kg, Part A (SAD) (N=6) | Investigational Drug, 0.6 mg/kg, Part A (SAD) (N=6) | Investigational Drug, 1.2 mg/kg, Part A (SAD) (N=6) | Placebo, Part A (SAD) (N=6) | Investigational Drug, 0.6 mg/kg, Part B (MAD) (N=8) | Investigational Drug, 1.2 mg/kg, Part B (MAD) (N=8) | Placebo, Part B (MAD) (N=4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Noninfective bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT05677893/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05677893/SAP_001.pdf